CLINICAL TRIAL: NCT07271030
Title: The Use of Cannabidiol Suppositories for Sexual Pain: A Randomised Controlled Study
Brief Title: The Use of Cannabidiol Suppositories for Sexual Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LondonsMUSB
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Well-Being, Psychological; Quality of Life; Sexual Behavior; Sexual Pain Disorder
MeSH Terms: conditions — Psychological Well-Being; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: The study phase is not applicable, as cannabidiol suppositories are not considered a drug.
  Randomisation would be based on dose specific groups, including, for example, 30, 50, 100mg and care as usual group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cannabidiol 30mg (Experimental): This will be a dose specific suppository of 30mg, which will be used for one month. Frequency will depend on how often the participant engages in sexual intimacy.
  Interventions: Dietary Supplement: Cannabidiol suppository intervention 1
- Cannabidiol 50mg (Experimental): This will be a dose specific suppository of 50mg, which will be used for one month. Frequency will depend on how often the participant engages in sexual intimacy.
  Interventions: Dietary Supplement: Cannabidiol suppository intervention 2
- Cannabidiol 100mg (Experimental): This will be a dose specific suppository of 100mg, which will be used for one month. Frequency will depend on how often the participant engages in sexual intimacy.
  Interventions: Dietary Supplement: Cannabidiol suppository intervention 3
- Care as usual (Active Comparator): This is the care as usual group, which will be the control for comparative outcomes with sexual function, sexual pain, well being and quality of life.
  Interventions: Other: Non cannabidiol group control

INTERVENTIONS:
Dietary Supplement: Cannabidiol suppository intervention 1 — Cannabidiol suppository dose specific 30mg
  Arms: Cannabidiol 30mg
Dietary Supplement: Cannabidiol suppository intervention 2 — Cannabidiol suppository dose specific 50mg
  Arms: Cannabidiol 50mg
Dietary Supplement: Cannabidiol suppository intervention 3 — Cannabidiol suppository dose specific 100mg
  Arms: Cannabidiol 100mg
Other: Non cannabidiol group control — Care as usual group
  Arms: Care as usual

SUMMARY:
Research aim: To determine how cannabidiol suppositories might reduce sexual pain during intimacy. Outcomes are also hoped to increase sexual functioning, well-being, and quality of life.

Research intention: If cannabidiol suppository intervention reduces sexual pain and increases general well-being, then this research would be repeated on a larger scale, targeting psychosexual services.

A brief overview of the intervention:

Quantitatively, randomisation of cannabidiol suppositories will be into dose-specific groups. The intervention will be delivered over a period of one month, with follow-up scheduled at 12 weeks. Qualitatively, participants were asked approximately eight open-ended feedback questions throughout the study.

DETAILED DESCRIPTION:
Sexual pain is a constellation of biopsychosocial disorders which affects men, women and their partners.

Cannabidiol is one of approximately 100 cannabinoids found in cannabis, alongside tetrahydrocannabinol. Cannabidiol is non-intoxicating and regarded as a safe product to use. Cannabidiol has many applications, including in sexual health. Two studies have examined cannabidiol suppositories for supporting sexual function and reducing sexual pain. In both studies, outcomes suggested the pain relieving qualities of cannabidiol oil for both men and women.

This research aims to establish the effectiveness of varied doses of cannabidiol oil to minimise sexual pain and increase well-being. This research is a preliminary study looking at how cannabidiol suppositories aim to reduce pain and support sexual function, wellbeing and quality of life among those experiencing sexual discomfort or pain during intercourse or masturbation.

There will be four groups, where cannabidiol will be randomised to dose-specific groups, approximately 30, 50, and 100mg, under the guidance of a medical practitioner. There will also be a care as usual group.

It is hypothesised that:

Higher levels of sexual functioning, quality of life and wellbeing with lower levels of sexual pain will be reported among those using cannabidiol suppositories at the follow-up after intervention compared to care as usual group.

It is further hypothesised that higher doses of cannabidiol suppositories will have higher levels of sexual pain-reducing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Has previously used cannabidiol in any capacity and has not experienced any allergic reaction
* Is experiencing sexual pain
* There will be an absence of co occurring difficulties
* Has attempted sexual intercourse in the last month
* Age 18 years or older
* Read and write English
* Patient Health Questionnaire 9 screening score range between 0-9 mild
* General Anxiety Disorder 7 screening score range between 0-9 mild
* There are no restrictions on sex, gender, sexuality, or disability

Exclusion Criteria:

Has experienced an allergic reaction to cannabidiol in any capacity

* Has not attempted sexual intercourse in the last month
* Has co occurring difficulties
* Aged below 18 years old
* Are not experiencing sexual pain
* Patient Health Questionnaire 9 screening score range between moderate to severe - 10-27
* General Anxiety Disorder 7 screening score range between 10- 21.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The Female Sexual Function Index | 0, 4 and 12 weeks
  This is a 19 item measure of sexual pain, sexual desire, orgasm, lubrication, and sexual satisfaction with five response categories. The score range is 2.0 to 36.0 with 26.0 being the cut of for sexual dysfunction. Example questions include, Over the past 4 weeks, how often did you experience discomfort or pain during vaginal penetration? and Over the past 4 weeks, how would you rate your level of discomfort or pain during or following vaginal penetration? Cronbach alpha for this questionnaire is .820 and higher.
The Short Warwick Edinburgh Mental Well-being Scale | 0, 4 and 12 weeks
  This is a 7 item questionnaire with 5 response categories looking at functioning and feeling aspects of well-being. The response categories include 1=none of the time to 5=all of the time. Cronbach alpha for the questionnaire is 0.89-0.91. There is no reverse scoring. Scores range from 7 to 35 where the latter is the highest level of wellbeing.
Brief Quality of Life Scale | Weeks 0, 4 and 12
  An 8 item questionnaire with five response categories looking at satisfaction with self, friends, family and creativity. This scale is scored by transforming the individual item scores from a 1 to 5 scale to a 0 to 100 scale. Example responses include how I view my life as necessary for my quality of life, and I am satisfied with my friends and friendship: The Cronbach alpha is .760 for this questionnaire
Changes in levels of anal pain taken | Weeks 0, 4 and 12
  The frequency and severity of pain during anal sex, this is a 5-point Likert-type scale which ranges from never (5) to all the time (1) and no anal pain (5) to severe anal pain (1). The Cronbach alpha in this study= 0.70.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Metropolitan University
Locations (1):
- School of Social Sciences and Professions, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitchell KR, Geary R, Graham CA, Datta J, Wellings K, Sonnenberg P, Field N, Nunns D, Bancroft J, Jones KG, Johnson AM, Mercer CH. Painful sex (dyspareunia) in women: prevalence and associated factors in a British population probability survey. BJOG. 2017 Oct;124(11):1689-1697. doi: 10.1111/1471-0528.14518. Epub 2017 Jan 25. PMID 28120373
- [Result] Nimbi FM, Rossi V, Tripodi F, Luria M, Flinchum M, Tambelli R, Simonelli C. Genital Pain and Sexual Functioning: Effects on Sexual Experience, Psychological Health, and Quality of Life. J Sex Med. 2020 Apr;17(4):771-783. doi: 10.1016/j.jsxm.2020.01.014. Epub 2020 Feb 13. PMID 32063471
- [Result] Lo LA, Christiansen AL, Strickland JC, Pistawka CA, Eadie L, Vandrey R, MacCallum CA. Does acute cannabidiol (CBD) use impair performance? A meta-analysis and comparison with placebo and delta-9-tetrahydrocannabinol (THC). Neuropsychopharmacology. 2024 Aug;49(9):1425-1436. doi: 10.1038/s41386-024-01847-w. Epub 2024 Mar 25. PMID 38528133
- [Result] Boardman LA, Stockdale CK. Sexual pain. Clin Obstet Gynecol. 2009 Dec;52(4):682-90. doi: 10.1097/GRF.0b013e3181bf4a7e. PMID 20393420
- [Result] Damon W, Rosser BR. Anodyspareunia in men who have sex with men: prevalence, predictors, consequences and the development of DSM diagnostic criteria. J Sex Marital Ther. 2005 Mar-Apr;31(2):129-41. doi: 10.1080/00926230590477989. PMID 15859372
- [Result] Haroutounian S, Ratz Y, Ginosar Y, Furmanov K, Saifi F, Meidan R, Davidson E. The Effect of Medicinal Cannabis on Pain and Quality-of-Life Outcomes in Chronic Pain: A Prospective Open-label Study. Clin J Pain. 2016 Dec;32(12):1036-1043. doi: 10.1097/AJP.0000000000000364. PMID 26889611
- [Result] Rosser BR, Short BJ, Thurmes PJ, Coleman E. Anodyspareunia, the unacknowledged sexual dysfunction: a validation study of painful receptive anal intercourse and its psychosexual concomitants in homosexual men. J Sex Marital Ther. 1998 Oct-Dec;24(4):281-92. doi: 10.1080/00926239808403963. PMID 9805288
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Banbury S, Tharmalingam H, Lusher J, Erridge S, Chandler C. A Preliminary Investigation into the Use of Cannabis Suppositories and Online Mindful Compassion for Improving Sexual Function Among Women Following Gynaecological Cancer Treatment. Medicina (Kaunas). 2024 Dec 7;60(12):2020. doi: 10.3390/medicina60122020. PMID 39768900
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Result] Lindner P, Frykheden O, Forsstrom D, Andersson E, Ljotsson B, Hedman E, Andersson G, Carlbring P. The Brunnsviken Brief Quality of Life Scale (BBQ): Development and Psychometric Evaluation. Cogn Behav Ther. 2016 Apr;45(3):182-95. doi: 10.1080/16506073.2016.1143526. Epub 2016 Feb 17. PMID 26886248